CLINICAL TRIAL: NCT02556749
Title: Effects of Cranberry Juice on Cardiovascular Risk Factors in a Placebo-controlled Crossover Trial
Brief Title: Effects of Cranberry Juice on Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Ocean Spray Cranberries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PKE CRAN
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease Risk Factors
Keywords: Cranberries; blood pressure; cholesterol; SphygmoCor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cranberry Juice Beverage (Experimental): 16 ounces of 54% cranberry juice cocktail
  Interventions: Dietary Supplement: Cranberry Juice Beverage
- Placebo Beverage (Placebo Comparator): Color, calorie, and taste matched beverage without cranberry bioactives
  Interventions: Dietary Supplement: Placebo Beverage

INTERVENTIONS:
Dietary Supplement: Cranberry Juice Beverage — 16 ounces of 54% cranberry juice cocktail
  Arms: Cranberry Juice Beverage
Dietary Supplement: Placebo Beverage — Color, calorie, and taste matched beverage without cranberry bioactives
  Arms: Placebo Beverage

SUMMARY:
The purpose of this study is to evaluate the effects of cranberry juice on central and peripheral blood pressure, indices of arterial stiffness, lipid and lipoprotein concentrations and size characteristics, and HDL function. The investigators hypothesize that the bioactive compounds in cranberry juice may elicit beneficial effects on blood pressure and arterial health, as well as LDL-C and HDL function.

DETAILED DESCRIPTION:
The investigators propose to conduct a 2-period randomized, crossover, placebo-controlled study to evaluate the effect of cranberry juice on central and peripheral blood pressure, indices of arterial stiffness, lipid and lipoprotein concentrations and size characteristics, and HDL function. Eligibility requires non-smoking men and women to be 30 to 65 years of age with BMI greater than or equal to 18 and less than or equal to 39, total cholesterol below 273 mg/dL for men and below 284 mg/dL for women, triglycerides below 350 mg/dL, and have systolic blood pressure of 120 to 159 mmHg and/or diastolic blood pressure of 80 to 99 mmHg. Subjects will undergo randomized treatments including 500 mL/d cranberry juice beverage and 500 mL/d of a color and taste matched placebo beverage. The two 8 to 12 week treatment periods will be separated by an 8 week washout.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 30-65 years of age
2. BMI ≥ 18 and ≤ 39 kg/m^2
3. Total cholesterol below 273 mg/dL for men and below 284 mg/dL for women
4. Triglycerides below 350 mg/dL
5. Non-smokers
6. At least one of the following:

   1. Systolic blood pressure 120-159 mmHg
   2. Diastolic blood pressure 80-99 mmHg

Exclusion Criteria:

1. History of acute or chronic inflammatory conditions or heart disease, kidney disease, liver disease, autoimmune disorders, or thyroid disease (unless controlled by medication and blood results within previous 6 months are provided)
2. History of diabetes mellitus (and/or a fasting glucose >126 mg/dL at screening)
3. Stage II hypertension (blood pressure ≥ 160/100 mmHg)
4. Lactation, pregnancy, or desire to become pregnant during the study
5. Unwillingness to discontinue nutritional supplements, herbs, or vitamins unless approved by investigator
6. Use of medications/supplements for elevated lipids, blood pressure, or glucose
7. Chronic use of non-steroidal anti-inflammatory or immunosuppressant medication
8. Conditions requiring the use of steroids
9. Unwillingness to refrain from blood donation prior to and during the study
10. Any medical condition or abnormal laboratory value that is judged clinically significant by an investigator
11. Allergy or sensitivity to cranberry juice or any ingredient in the study beverages

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-10; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Central Blood Pressure | Change from baseline after 8 week treatments with cranberry and placebo
  Aortic (central) blood pressure measured using the SphygmoCor system
Peripheral Blood Pressure | Change from baseline after 8 week treatments with cranberry and placebo
  Peripheral blood pressure measured using the SphygmoCor system

SECONDARY OUTCOMES:
Efflux capacity of HDL | Change from baseline after 8 week treatments with cranberry and placebo
  Ability to carry out reverse cholesterol transport measured using in vitro assay
Augmentation Index | Change from baseline after 8 week treatments with cranberry and placebo
  Augmentation index measured using the SphygmoCor system
Pulse Wave Velocity | Change from baseline after 8 week treatments with cranberry and placebo
  Pulse wave velocity measured using the SphygmoCor system
LDL-C | Change from baseline after 8 week treatments with cranberry and placebo
  LDL-C values calculated using the Friedewald equation
LDL Particle Size | Change from baseline after 8 week treatments with cranberry and placebo
  LDL particle size measured using a Vertical Auto Profile (VAP) Test
Total Cholesterol | Change from baseline after 8 week treatments with cranberry and placebo
  Total cholesterol values determined by enzymatic procedures
Triglycerides | Change from baseline after 8 week treatments with cranberry and placebo
  Triglyceride values determined using enzymatic procedures
HDL-C | Change from baseline after 8 week treatments with cranberry and placebo
  HDL-C will be estimated according to the modified heparin-manganese procedure
Oxidized LDL (oxLDL) | Change from baseline after 8 week treatments with cranberry and placebo
  Plasma concentrations of oxLDL will be measured using ELISA kits
Malondialdehyde (MDA) | Change from baseline after 8 week treatments with cranberry and placebo
  MDA will be measured using the thiobarbituric acid reactive substances (TBARS) assay
High Sensitivity C Reactive Protein (hs-CRP) | Change from baseline after 8 week treatments with cranberry and placebo
  hs-CRP will be measured by latex-enhanced immunonephelometry
24-hr Ambulatory Blood Pressure | Change from baseline after 8 week treatments with cranberry and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Penny Kris-Etherton, PhD, RD, Principal Investigator — Penn State University
Locations (1):
- Penn State CRC, University Park, Pennsylvania, United States